CLINICAL TRIAL: NCT03671681
Title: A Randomized Clinical Trial on the Efficacy and Cost-efficacy of Adding on a Mindfulness-based Therapy to Standard Medical Prophylaxis in the Treatment of Patients With Chronic Migraine Associated to Medication Overuse Following Structured Withdrawal: the Mind-CM Study
Brief Title: Mindfulness Therapy for Chronic Migraine
Acronym: Mind-CM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mind-CM
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Chronic Migraine; Medication Overuse Headache
Keywords: Chronic Migraine; Medication Overuse Headache; Mindfulness; Pharmacological Prophylaxis; Neuroimaging; Neuroinflammation; Disability; Quality of Life; Depression; Anxiety
MeSH Terms: conditions — Headache Disorders, Secondary; Neuroinflammatory Diseases; Depression; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MT group (Experimental): Education of patients, Pharmacological Prophylaxis prescribed based on patients' profile, and six group sessions of 45 minutes of mindfulness-based treatment.
  Interventions: Behavioral: Mindfulness; Drug: Prophylactic
- MED group (Other): Education of patients followed by Pharmacological Prophylaxis, prescribed based on patients' profile (i.e. clinical features, previous failures and contraindications)
  Interventions: Drug: Prophylactic

INTERVENTIONS:
Behavioral: Mindfulness — The experimental group will receive education, will be prescribed prophylaxis and will attend Mindfulness-based therapy sessions. The MINDFULNESS therapy consists in 6 weekly sessions, 45 minutes each. The main focus of the six mindfulness session will be the following: 1) introduction and meaning; 2) Focus on breath; 3) posture and body awareness; 4) meditation of sounds; 5) Guided imagery; 6) acceptance and awareness. During training, patients will be invited to close their eyes, assume a relaxed position, focus on their breathing and on the present to enhance awareness of current mind and body sensations. Patients will be trained in small groups (5-7 patients each) and guided by a specifically trained therapist. They will be educated to practice at home according to the instructions given by the therapist during the sessions.
  Arms: MT group
Drug: Prophylactic — Control group will receive education on the use of pharmacological compounds for acute treatment and on healthy lifestyle habits (e.g. adequate sleep/wake pattern, eating and hydration, physical activity, avoidance of triggers) and will be prescribed prophylactic medications. The preventive compound will be chosen on the basis of clinical profile among the following categories: neuromodulators (e.g. topiramate or valproate), antidepressant (e.g. tricyclics or SSRIs) or others, e.g. beta-blockers.

SUMMARY:
The aim is to assess the efficacy of adding on a Mindfulness-based therapy to pharmacological prophylaxis (experimental group: pharmacological prophylaxis + Mindfulness) against pharmacological prophylaxis only (control group) on the reduction of monthly headaches frequency (primary endpoint), symptomatic medications intake, inflammatory pattern, depression, anxiety, cutaneous allodynia, improving disability and quality of life (secondary endpoints). Moreover, other aims are to assess whether adding on Mindfulness-based therapy is also associated to a superior improvement of neuroimaging pattern among patients prescribed neuromodulators or antidepressants and to assess the cost-efficacy of adding on a Mindfulness-based therapy to pharmacological prophylaxis. Mindfulness will be provided in small groups (5-7 patients each) by specifically trained therapists. The treatment consists in six 45 minutes weekly sessions in which one will work on meditation, acceptance and awareness. The program of control group will consist in education of patients, followed by pharmacological prophylaxis. Prophylaxis is prescribed based on patients' profile, such as previous failures, contraindications and so on by a neurologist with expertise in headache treatments. We expect that adding-on Mindfulness will determine a wider reduction of headaches frequency and improvement of secondary endpoints, and that disease cost reduction will support the cost-efficacy of Mindfulness. The study will be a Phase III; randomized, Open-Label; Monocentric study. Patients will be enrolled to detect a 20% difference between the two groups on the primary outcome (50% or more of headache reduction by 12 months). For each medication type and research arm 20 patients will be selected: thus 80 patients will be enrolled for neuroradiological investigation.

DETAILED DESCRIPTION:
Background and significance. Chronic migraine (CM) is a negative evolution of migraine characterized by frequent headache attacks (>45 days/three months) with a 1-year prevalence of 3.1%. Comorbidities, lifestyle and excessive intakes of symptomatic medications (medication overuse-MO) play a role in progression into CM; altered inflammatory state (WBC, peripheral blood lymphocyte subsets CD3, CD4, CD8, CD19) and dysfunctions in the mesocorticolimbic dopamine circuit were found in CMMO patients. To prevent CM-MO relapse, withdrawal of overused drugs and complementing pharmacological prophylaxis with behavioral treatments is indicated [5]. Withdrawal from MO and medical prophylaxis determine a 30-40% reduction in headaches frequency by 12 months, and 40-50% of patients show a reduction >=50%. Conversely, 30% of them relapse into CM-MO by 12 months: the main drivers include overuse of analgesic compared to triptans and being on medical therapy alone compared to adjuvant psychological techniques. Research demonstrated the utility of relaxation training, stress management, cognitive-behavioral therapy in migraine disorder. Parallel to this, mindfulness showed considerable promise particularly on headache-related disability, affective distress: however, to date evidence of its efficacy is limited by small trials, short follow-up periods, inadequate power and poor consideration of primary outcomes for CM research, i.e. reduction of headaches frequency. Our main hypothesis is that mindfulness might provide additional benefit, when added to medical prophylaxis alone, on both primary (i.e. an increased number of patients showing a reduction of headaches frequency >=50%) and secondary outcomes: reduction in the consumption of symptomatic medications (i.e. analgesics, triptans, opioids, ergot-derivate), reduction of disability, depression, anxiety and cutaneous allodynia, improvement in quality of life; reduction of costs, connected to both lower direct medical costs (e.g. drugs consumption and attendance to ER) and indirect costs (i.e. reduction in lost workdays and improved workplace efficiency); reduction in concentration of the markers of inflammatory pattern; reversible neuroadaptations highlighted by functional connectivity in regions of dopaminergic circuit.

The study will be a Phase III; randomized, Open-Label; Monocentric study. Patients will be enrolled to detect a 20% difference between the two groups on the primary outcome (50% or more of headache reduction by 12 months). We set alpha 0.05 and power 80%, and foresee that up to 12% of patients might be lost at follow-up: therefore, we determined that 170 patients should be randomized 1:1 to the two groups. Patients will be excluded if they: have psychiatric comorbidities of psychotic area; pregnancy; comorbidity with secondary headaches (e.g. idiopathic intracranial hypertension); were submitted to withdrawal from MO at least twice in the previous two years; attended any mindfulness-based therapy. For each medication type and research arm 20 patients will be selected: thus 80 patients will be enrolled for neuroradiological investigation. The treatment consists in six 45 minutes weekly sessions. The main focus of the six session will be the following: 1) introduction and meaning; 2) Focus on breath; 3) posture and body awareness; 4) meditation of sounds; 5) Guided imagery; 6) acceptance and awareness.

Our project is highly innovative as it will be the first time in which a new emerging treatment like Mindfulness is tested for its efficacy and cost-efficacy when added to standard pharmacological prophylaxis. If our hypothesis will be confirmed, then we will positively impact on: a) clinicians, that will have confirmation of another valid adjuvant treatment option; b) national health system, that will cut down the relevant costs of medication intake and indirect costs associated to reduced productivity; c) patients, that will enhance their ability to cope with headaches and improve their overall health, quality of life, work-ability and reduce their disability. Moreover, our study will address the possible impact of Mindfulness as an add-on to pharmacological prophylaxis not only on clinical data, such as headaches frequency and symptomatic medications intake, but also on biomarkers of inflammatory and functional neuroimaging patterns.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Migraine (migraine headaches on ≥15 days of migraine headache per month, for three consecutive months) associated to Medication overuse (Regular intake for >3 months of analgesics on >=15 days/month or of triptans, ergotamine, NSAID, opioids or multiple drugs on >=10 days/month). Diagnoses are made according to the third version of the International Classification of Headache Disorders (code 1.3-Chronic Migraine; code 8.2-Medication Overuse Headache).

Exclusion Criteria:

* psychiatric comorbidities of psychotic area;
* pregnancy;
* comorbidity with secondary headaches (e.g. idiopathic intracranial hypertension);
* submitted to withdrawal from MO at least twice in the previous two years;
* attended any mindfulness-based therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Headache frequency reduction | 12 months
  Percentage of patients achieving 50% or more of headache frequency reduction at 12-months compared to baseline assessed with headache diary.

SECONDARY OUTCOMES:
Neuroimaging pattern | 12 months
  Change in neuroimaging pattern among patients prescribed neuromodulators (e.g. valproate or topiramate) or antidepressants (e.g. tricyclics or SSRIs) assessed with functional magnetic imaging (rs-fMRI).
Cost-efficacy | 3, 6, 12 months
  Differences in cost-efficacy of adding on a Mindfulness-based therapy to pharmacological prophylaxis assessed with self-reports in which patients specify lost workdays and days worked with reduced efficacy (indirect costs), and drug intake by type and medical procedures (direct costs).
Health and disability | 3, 6, 12 months
  Change in health and disability scores, assessed with the WHO Disability Assessment Schedule 2.1 (WHODAS 2.0) WHODAS 2.0 covers 6 Domains of Functioning, including: Cognition, Mobility, Self-care, Getting along , Life activities, Participation. Each item has 5 answers with their scores from "none" to "extreme". The summary score ranges from 0-100 (0 = no disability; 100 = full disability).
Disability | 3, 6, 12 months
  Change in disability scores, assessed with Headache Impact Test-6 (HIT-6) The HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The patient answers each of the six related questions using one of the following five responses: "never", "rarely", "sometimes", "very often", or "always". Each answer is associated with a different score: "never" 6 points, "rarely" 8 points, "sometimes" 10 points, "very often" 10 points," always" 13 points. These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent.
Change in Quality of life | 3, 6, 12 months
  Change in quality of life, assessed with the Migraine-Specific Quality of Life Questionnaire 2.1 (MSQ 2.1) The MSQ is a 14-item instrument that measures the impact of migraine across three essential aspects of a patient's health-related quality of life over the past 4 weeks: role function-restrictive (7 items assessing how migraines limit one's daily social and work-related activities) , role function-preventive (4 items assessing how migraines prevent these activities), and emotional function (3 items assessing the emotions associated with migraines). Participant respond to items using a 6-point scale: "none of the time," "a little bit of the time," "some of the time," "a good bit of the time," "most of the time," and "all of the time," which are assigned scores of 1 to 6, respectively. Raw dimension scores are computed as a sum of item responses and rescaled from a 0 to 100 scale such that higher scores indicate better quality of life.
Depression | 3, 6, 12 months
  Change in depression scores, assessed with beck depression inventory-II and (BDI-II) The BDI-II is a questionnaire composed of 21 items that refer to a wide range of somatic affective and cognitive symptoms related to depression. For each item the subject must respond by choosing between 4 alternatives corresponding to different levels of severity. Each alternative is associated with a score ranging from 0 to 3. Total score is obtained by adding the scores of each item. The total score ranges from 0 to 63. Higher scores indicate more severe depressive symptoms: 0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, 29-63: severe depression.
Anxiety | 3, 6 and 12 months
  Change in anxiety scores, assessed with state-trait anxiety inventory forme Y (STAY-Y) STAI comprises separate self-report scales for measuring state and trait anxiety.
  STAI comprises separate self-report scales for measuring state and trait anxiety. The STAI Form Y-1 consists of 20 statements that evaluate how respondents feel "right now, at this moment". The STAI Form Y-2 consists of 20 statements that assess how people generally feel. Each STAI item is given a weighted score of 1 to 4. Scores for both can vary from a min of 20 to a max of 80.
Allodynia | 3, 6 and 12 months
  Change in allodynia, assessed with the Allodynia Symptom Checklist (ASC)
Inflammatory pattern | 6 and 12 months
  Change in Biomarkers of inflammatory pattern (WBC, lymphocyte subsets CD3, CD4, CD8, CD19, Treg cells, IL6) The units of measurement, WBC and lymphocyte subpopulations (CD3, CD4, CD8, CD19, Treg), are expressed in number / ml, IL-6 in pg / mL. The different parameters are not aggregated for a composite measure.
Medications consumption | 3, 6 and 12 months
  Change in medications consumption assessed with headache diary

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Neuroalgology Unit, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Scientific conferences, publications

REFERENCES:
- [Derived] Grazzi L, D'Amico D, Guastafierro E, Demichelis G, Erbetta A, Fedeli D, Nigri A, Ciusani E, Barbara C, Raggi A. Efficacy of mindfulness added to treatment as usual in patients with chronic migraine and medication overuse headache: a phase-III single-blind randomized-controlled trial (the MIND-CM study). J Headache Pain. 2023 Jul 14;24(1):86. doi: 10.1186/s10194-023-01630-0. PMID 37452281
- [Derived] Grazzi L, Raggi A, Guastafierro E, Passavanti M, Marcassoli A, Montisano DA, D'Amico D. A Preliminary Analysis on the Feasibility and Short-Term Efficacy of a Phase-III RCT on Mindfulness Added to Treatment as Usual for Patients with Chronic Migraine and Medication Overuse Headache. Int J Environ Res Public Health. 2022 Oct 29;19(21):14116. doi: 10.3390/ijerph192114116. PMID 36360996